CLINICAL TRIAL: NCT04085393
Title: Granisetron Extended Release Injection (GERSC) for the Prevention of Chemotherapy-induced Breakthrough Nausea and Vomiting (CINV) in Patients Receiving Moderately or Highly Emetogenic Chemotherapy: A Phase II Clinical Trial
Brief Title: Granisetron Extended Release Injection (GERSC) for the Prevention of Chemotherapy-induced Nausea and Vomiting
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor withdrew study
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Heron Therapeutics (Industry)
Responsible Party: Principal Investigator, Rudolph Navari, Professro, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAB1950
Record Dates: First submitted 2019-08-29; First posted 2019-09-11 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GERSC for patients receiving highly emetogenic chemotherapy (Active Comparator): Participants will receive GERSC, and two other standard antiemetics prior to chemotherapy
  Interventions: Drug: GRANISETRON EXTENDED RELEASE INJECTION (GERSC)
- GERSC on patients receiving moderately emetogenic chemotherapy (Active Comparator): Participants will receive GERSC and one other standard antiemetic prior to chemotherapy
  Interventions: Drug: GRANISETRON EXTENDED RELEASE INJECTION (GERSC)

INTERVENTIONS:
Drug: GRANISETRON EXTENDED RELEASE INJECTION (GERSC) — GERSC is a new, subcutaneously (SC) administered polymeric formulation of granisetron that was developed to provide slow, controlled, and sustained release of granisetron to prevent both acute and delayed CINV associated with MEC and HEC. Due to the prolonged efficacy, GERSC may potentially improve CINV in the acute and delayed periods and the single dose regimen may improve patient adherence to antiemetic therapy

SUMMARY:
Chemotherapy-induced nausea and vomiting (CINV) adversely affects patients' quality of life and may affect patients' treatment decisions. The emetogenicity of the chemotherapy administered and specific patient characteristics such as female gender, age, and history of low alcohol intake can increase a patients' risk for CINV.

GERSC is a new, subcutaneously (SC) administered polymeric formulation of Granisetron that was developed to provide slow, controlled, and sustained release of Granisetron to prevent both acute and delayed CINV associated with moderately emetic chemotherapy (MEC) and highly emetic chemotherapy (HEC)

DETAILED DESCRIPTION:
All patients eligible for the study receiving moderately emetogenic (MEC) chemotherapy will receive GERSC receptor antagonist on day one. All patients eligible for the study receiving highly emetogenic Chemotherapy (HEC) chemotherapy will receive GERSC receptor antagonist on day one including dexamethasone and NK-1 Receptor antagonist during cycle 1.

The primary objective is to measure the Complete Response (no emetic episodes, no use of rescue medications) in patients receiving GERSC as a replacement for the second generation 5 HT3 receptor antagonist palonosetron used in the first chemotherapy cycle for those patients receiving MEC or HEC and developed Breakthrough CINV. Complete response would be recorded specifically for the acute (0-24 hours post-chemotherapy), delayed (24-120 hours post-chemotherapy), and overall periods (0-120 hours post-chemotherapy).

This study has two study groups.

* Group 1 (HEC) will receive GERSC, dexamethasone and NK-1 antagonist prior to chemotherapy
* Group 2 (MEC) will receive GERSC and dexamethasone prior to chemotherapy

During the study:

Participants will be completing questionnaires on day 1 prior to treatment and at approximately the same time treatment was given each day for the next seven days. Participant will be assessed each day on the amount of nausea, vomiting, and/or sedation experienced in the previous 24-hour period. The assessment should take less than 5 minutes to complete each day.

Participants will be registered for Quality of Life measurement. Validated QOL measurements of fatigue and overall perception of QOL will be assessed upon registration in this study. Fatigue and overall well-being clearly can impact how well patients will do in terms of being able to tolerate and experience nausea and vomiting

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignant disease and scheduled for MEC or HEC
* Chemotherapy naive
* Age ≥18 years.
* ECOG Performance Status 0 or 1
* Required Initial Laboratory Values ≤28 days prior to registration. Patient must have adequate bone marrow, kidney, and liver function as evidenced by:
* Platelet count ≥ 100,000/ mm3
* Bilirubin ≤ 1.5 x ULN, except for subjects with Gilbert's syndrome
* Serum Creatinine ≤2.0 mg/dL
* SGOT or SGPT ≤3 x upper limit of normal (ULN)
* Absolute neutrophil count (ANC) ≥1500/mm3
* Patients receiving HEC will have received the 5HT3 receptor antagonist palonosetron, a NK-1, and dexamethasone as antiemetic prophylaxis during cycle 1 of chemotherapy
* Patients receiving MEC will have received the 5HT3 receptor antagonist palonosetron, and dexamethasone as antiemetic prophylaxis during cycle 1 of chemotherapy

Exclusion Criteria:

* No nausea or vomiting ≤ 24 hours prior to registration.
* Negative pregnancy test (serum β hCG) done ≤7 days prior to registration, for women of childbearing potential only (per clinician discretion).
* No severe cognitive compromise.
* No known history of active, untreated CNS disease (e.g. brain metastases, seizure disorder).
* No concurrent use of amifostine, thioridazine, pimozide or St. John's wort.
* No concurrent abdominal radiotherapy.
* No concurrent use of olanzapine therapy.
* No chronic alcoholism (as determined by the investigator).
* No known hypersensitivity to granisetron.
* No known uncontrolled cardiac arrhythmia or uncontrolled congestive heart failure.
* No acute myocardial infarction within the previous six months.
* No history of uncontrolled diabetes mellitus (may be on a stable dose of insulin or on a stable dose of an oral hypoglycemic agent).
* Patients with psychiatric illness that would prevent the patient from giving informed consent are not eligible for the trial
* Medical condition such as uncontrolled infection (including HIV),uncontrolled Diabetes Mellitus, unstable cardiac disease which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient are not eligible for the trial
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers are not eligible for the trial; Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 3 years.
* Patients who cannot swallow oral formulations of the agent(s) are not eligible for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with a previous history of emetic episodes | Baseline assessment
  After participants have completed their informed consent, they will complete a baseline assessment to record emetic episodes prior to chemotherapy.
Percentage of participants with a complete response of no emetic episode | Baseline through 24 hours
  Patient will be monitored for vomiting on Day 1 after receiving chemotherapy. The participants will complete a vomiting assessment and record the number of episodes (none, once, more than once and number)
Percentage of participants with a complete response of no emetic episode | Day 2 through Day 6
  Patient will be monitored for vomiting on Day 2 through Day 6 after receiving chemotherapy. The participants will complete a vomiting assessment and record the number of episodes (none, once, more than once and number)
Percentage of participants with a complete response of no emetic episode | Day 1 through Day 6
  Patient will be monitored for total vomiting episodes starting from Day 1 through Day 6 after receiving chemotherapy. The participants will complete a vomiting assessment and record the number of episodes (none, once, more than once and number)

SECONDARY OUTCOMES:
Percentage of participants frequency rate of No Nausea | Baseline
  Participants will complete a Visual Analogue Scale at baseline to record their history of the presence or absence of nausea and frequency prior to chemotherapy. The scale range is between 0 - 10 (0 = No Nausea; 10 = Excessive Nausea).
Percentage of participants frequency rate of No Nausea | Baseline through 24 hours
  Participants will complete a Visual Analogue Scale on Day 1 to record the presence or absence of nausea and frequency after receiving chemotherapy. The scale range is between 0 - 10 (0 = No Nausea; 10 = Excessive Nausea).
Percentage of participants frequency rate of No Nausea | Day 2 through Day 6
  Participants will complete a Visual Analogue Scale on Day 2 through Day 6 to record the presence or absence of nausea and frequency after receiving chemotherapy. The scale range is between 0 - 10 (0 = No Nausea; 10 = Excessive Nausea).
Percentage of participants frequency rate of No Nausea | Day 1 through Day 6
  Participants will complete a Visual Analogue Scale on Day 1 through Day 6 to record the presence or absence of nausea and frequency after receiving chemotherapy. The scale range is between 0 - 10 (0 = No Nausea; 10 = Excessive Nausea).
Percentage of participants experiencing GERSC toxicity | Baseline through 30 days
  The toxicity will be assessed by the severity of the side effects listed below. The descriptions and grading scales found in the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 will be utilized for reporting.
  * Constipation
  * Fatigue
  * Headache
  * Diarrhea
  * Abdominal Pain
  * Sleeplessness (Insomnia)
  * Indigestion (Dyspepsia)
  * Dizziness
  * Asthenia
  * Gastroesophageal Reflux

CONTACTS AND LOCATIONS:
Overall Officials: Rudolph M Navari, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No